CLINICAL TRIAL: NCT06743776
Title: Scalable Expanded Access With Analysis of Neurofilament and Other Biomarkers for Ibudilast in ALS
Acronym: SEANOBI-ALS
Status: Available | Type: Expanded Access
Sponsor: Mayo Clinic (Other)
Collaborators: WideTrial, Inc. (Industry); MediciNova (Industry); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Bjorn E. Oskarsson, Associate Professor of Neurology, Mayo Clinic
Other Study IDs: 24-009898; U01NS136022 (NIH)
Record Dates: First submitted 2024-11-20; First posted 2024-12-20 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: ALS
MeSH Terms: interventions — ibudilast

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: MN-166 — MN-166 will be taken orally at a dose of 10 mg in the morning and 20 mg in the evening for the first 2 weeks, whereafter dose of 30 mg BID will be taken.

SUMMARY:
The purpose of this Expanded Access Program is to provide MN-166 (ibudilast) to ALS patients who are not eligible for an enrolling ALS clinical trial. This Expanded Access Program will assess if MN-166 can help people with ALS in slowing down the progression of the disease.

ELIGIBILITY:
Inclusion Criteria

1. ALS by "Gold Coast" diagnostic criteria
2. Age > 18 years
3. Either I) Ineligibility for interventional ALS clinical research participation due to at least one of the following standard exclusion criteria:

   1. Time since onset of weakness due to ALS > 36 months
   2. Vital Capacity less than 50% of predicted capacity for age, height, and sex measured (by Slow Vital Capacity (SVC) or Forced Vital Capacity (FVC))
   3. Cancer or history of cancer, except for the following: basal cell carcinoma or successfully treated squamous cell carcinoma of the skin, cervical carcinoma in situ, prostatic carcinoma in situ, or other malignancies curatively treated and with no evidence of disease recurrence for at least 3 years.
   4. Geographic inaccessibility from nearest actively enrolling research trial site for a trial the patient would otherwise qualify for, defined as either >200 miles or, in the opinion of the investigator, a distance that would make trial participation infeasible for the particular patient, due to significant disease progression or special logistical circumstances. OR II) Former COMBAT-ALS participant or current participant who has completed dosing in the OLE and may be consented at the final OLE follow-up visit.
4. Female patients of childbearing potential must use one or more effective methods of contraception throughout the entire EAP and for 30 days after discontinuing MN-166.
5. Male patients agree to practice contraception (e.g., condom use and contraception by female partner) unless partner is post-menopausal or unable to conceive throughout the entire EAP and for 30 days after discontinuing MN-166.

Exclusion Criteria

1. Clinically significant unstable medical condition (other than ALS) that would pose a risk to the participant, according to treating physician's judgment (e.g., psychiatric, cardiovascular instability, systemic infection, untreated thyroid dysfunction, or clinically significant laboratory abnormality or ECG changes).
2. Clinically significant lab abnormalities in the opinion of the treating physician, including, but not limited to: alanine aminotransferase (ALT) or aspartate aminotransferase (AST) or total bilirubin greater than 3 times the upper limit of normal (ULN), white blood cell count <2500/mm3, platelet count <75,000/mm3
3. Active drug or alcohol abuse
4. Female patient is lactating, pregnant, or planning pregnancy at Clinical Screening or Lab Screening
5. Concomitant use of another investigational medical product for treatment of ALS. Any such investigational medical product must be discontinued for a minimum of 5 half-lives prior to the first dose of MN-166.
6. Concomitant use of prohibited medications. Refer to Program Procedure Manual Appendix 3 for a list of prohibited medications.
7. Past participant in COMBAT-ALS clinical trial who did not complete the study.
8. Past participant in an ALS research trial who did not complete the study without cause.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Bjorn E Oskarsson, MD, Principal Investigator — Mayo Clinic
Locations (14):
- United States (14):
  - Mayo Clinic, Scottsdale, Arizona
  - University of California, San Francisco, San Francisco, California
  - Hospital for Special Care, New Britain, Connecticut
  - Nova Southeastern University, Davie, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Augusta University, Augusta, Georgia
  - Indiana University - IU Health Neuroscience Center, Indianapolis, Indiana
  - Hennepin Healthcare Research Institute, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - SUNY Upstate Medical University, Syracuse, New York
  - Duke University, Durham, North Carolina
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - Semmes Murphey Foundation, Memphis, Tennessee
  - University of Virginia, Charlottesville, Virginia